CLINICAL TRIAL: NCT00005940
Title: Phase II Study of Radiolabeled BC8 (Anti-CD45) Antibody Combined With Busulfan and Cyclophosphamide as Treatment for Acute Myelogenous Leukemia in First Remission Followed by HLA-Identical Related Peripheral Blood Stem Cell Transplantation
Brief Title: Radiolabeled BC8 Antibody, Busulfan, Cyclophosphamide Followed by Donor Stem Cell Transplant in Treating Patients With Acute Myelogenous Leukemia in First Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1470.00; NCI-2013-01361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHCRC-1470.00; NCI-H00-0056; 1470; CDR0000067778; 1470.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA044991 (NIH)
Record Dates: First submitted 2000-07-05; First posted 2003-07-09 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22)
MeSH Terms: conditions — Congenital Abnormalities | interventions — Busulfan; Cyclophosphamide; Transplantation; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (radiolabeled BC8, chemotherapy, PBSCT) (Experimental): RADIOLABELED ANTIBODY: Patients receive iodine I 131 monoclonal antibody BC8 IV on day -13.
  CHEMOTHERAPY: Patients receive busulfan PO every 6 hours on days -7 to -4 and cyclophosphamide IV on days -3 and -2.
  TRANSPLANT: Patients undergo allogeneic PBSC or BM transplant on day 0.
  GRAFT-VS-HOST DISEASE PREVENTION: Patients receive cyclosporine IV or PO every 12 hours on days -1 to 50 with a taper to day 180. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Radiation: iodine I 131 monoclonal antibody BC8; Drug: busulfan; Drug: cyclophosphamide; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: methotrexate; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody BC8 — Given IV
  Other Names: I 131 MOAB BC8; I 131 Monoclonal Antibody BC8; iodine I 131 MOAB BC8
Drug: busulfan — Given PO
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Procedure: allogeneic bone marrow transplantation — Undergo allogeneic PBSC or bone marrow transplant
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSC or bone marrow transplant
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic PBSC or bone marrow transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: cyclosporine — Given IV or PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well iodine I 131 monoclonal antibody BC8, busulfan, and cyclophosphamide followed by donor stem cell transplant works in treating patients with acute myeloid leukemia that has decreased or disappeared, but the cancer may still be in the body. Giving chemotherapy drugs, such as busulfan and cyclophosphamide before a donor peripheral blood stem cell transplant helps stop the growth of cancer or abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. Also, radiolabeled monoclonal antibodies, such as iodine I 131 monoclonal antibody BC8, can find cancer cells and carry cancer-killing substances to them without harming normal cells. When the stem cells from a related donor, that closely matches the patient's blood, are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy (as measured by survival and disease-free survival) and toxicity of a regimen of busulfan 16 mg/kg and cyclophosphamide 120 mg/kg plus 131I-labeled anti-cluster of differentiation (CD) 45 antibody (iodine I 131 monoclonal antibody BC8) (delivering a dose of 5.25 gray [Gy] to the normal organ receiving the highest dose) in patients with acute myeloid leukemia (AML) in first remission receiving human leukocyte antigen (HLA)-identical related peripheral blood stem cell (PBSC) transplants.

OUTLINE:

RADIOLABELED ANTIBODY: Patients receive iodine I 131 monoclonal antibody BC8 intravenously (IV) on day -13.

CHEMOTHERAPY: Patients receive busulfan orally (PO) every 6 hours on days -7 to -4 and cyclophosphamide IV on days -3 and -2.

TRANSPLANT: Patients undergo allogeneic PBSC or bone marrow (BM) transplant on day 0.

GRAFT-VS-HOST DISEASE PREVENTION: Patients receive cyclosporine IV or PO every 12 hours on days -1 to 50 with a taper to day 180. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed up at 6, 9, and 12 months; every 6 months for 1 year; and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML in first remission
* Creatinine < 2.0 mg/dl
* Bilirubin < 1.5 mg/dl which is expected to exclude patients at high risk of developing veno-occlusive disease of the liver
* Aspartate aminotransferase (AST) < 1.5 times the upper limit of normal which is expected to exclude patients at high risk of developing veno-occlusive disease of the liver
* Patients must have an expected survival of > 60 days and must be free of major infection
* DONOR: genotypic or phenotypic HLA-matched family members; related donors should be matched by molecular methods at the intermediate resolution level at HLA-A, B, C, and DR beta 1 (DRB1) according to Fred Hutchinson Cancer Research Center (FHCRC) Standard Practice Guidelines and to the allele level at DQ beta 1 (DQB1)

Exclusion Criteria:

* Patients with history of or current leukemic involvement of the central nervous system (CNS)
* Prior radiation to maximally tolerated levels to any normal organ
* Inability to understand or give an informed consent
* Patients who are seropositive for human immunodeficiency virus (HIV)
* Perceived inability to tolerate diagnostic or therapeutic procedures, particularly treatment in radiation isolation
* Circulating antibody against mouse immunoglobulin
* DONOR: unrelated donors and donors mismatched for 1 or more HLA antigens
* DONOR: donors who for psychologic, physiologic or medical reasons are unable to undergo filgrastim (G-CSF)- mobilized PBSC collection or marrow harvesting
* DONOR: donors who are seropositive for HIV

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 1999-10; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Up to 6 years
  Summarized using appropriate time-to-event methods with estimates of the corresponding confidence intervals provided.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 6 years
  Summarized using appropriate time-to-event methods with estimates of the corresponding confidence intervals provided.
Relapse of AML patients | Up to 6 years
  Summarized using appropriate time-to-event methods with estimates of the corresponding confidence intervals provided.
Transplant-related mortality | Up to 6 years
  Transplant-related toxicities are graded using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 2. Summarized using appropriate time-to-event methods with estimates of the corresponding confidence intervals provided.

CONTACTS AND LOCATIONS:
Overall Officials: Johnnie Orozco, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Pacific Northwest National Laboratory, Richland, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington